CLINICAL TRIAL: NCT02546297
Title: The Comparisons of the Efficacy and Safety of Inhaled LAMA or LAMA+LABA or ICS+LABA for Patients in COPD C Group With Bronchiectasis
Brief Title: Comparisons of Inhaled LAMA or LAMA+LABA or ICS+LABA for COPD With Bronchiectasis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Jin-Fu Xu, Department of Respiratory Medicine, Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20150717
Record Dates: First submitted 2015-07-22; First posted 2015-09-10 (Estimated); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: COPD; Bronchiectasis
Keywords: LAMA,ICS+LABA,LAMA+LABA
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchiectasis | interventions — Budesonide, Formoterol Fumarate Drug Combination; Tiotropium Bromide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- ICS/LABA Group (Active Comparator): Symbicort，Inhalation，Individualized medication，12 months.
  Interventions: Drug: Symbicort
- LAMA Group (Active Comparator): Tiotropium Bromide，Inhalation,Individualized medication，12 months.
  Interventions: Drug: Spiriva
- LAMA+LABA Group (Active Comparator): Tiotropium Bromide, Symbicort, Inhalation, Individualized medication, 12 months.
  Interventions: Drug: Symbicort; Drug: Spiriva

INTERVENTIONS:
Drug: Symbicort — drug are used for 12 months
  Other Names: Budesonide/Formoterol
  Arms: ICS/LABA Group; LAMA+LABA Group
Drug: Spiriva — drug are used for 12 months
  Other Names: Tiotropium Bromide
  Arms: LAMA Group; LAMA+LABA Group

SUMMARY:
The purpose of this study is to determine which treatment is more effective and safer for the patients in COPD C group with bronchiectasis.The research results will help guide physicians to select appropriate individualized treatment and hopefully provide some evidence-based medicine proofs for revising guide.

DETAILED DESCRIPTION:
The diagnosis and treatment of COPD and bronchiectasis together seems to be more complicated than the diagnosis and treatment of either condition alone. According to the GOLD，there are three treatments for patients with COPD in group C: ICS combined with LABA or LAMA alone or LABA combined with LAMA. However, it has not yet been demonstrated about which method is more effective for the patients with COPD in group C and bronchiectasis.

This study is designed as a prospective, randomized, case-control trial. Patients are divided into three groups, one group inhaled with ICS and LABA (Symbicort), the second group inhaled with LAMA (Tiotropium Bromide) and the third group inhaled with LAMA(Tiotropium Bromide) and (Symbicort).The course of treatment is 12 months.

The investigators will also assess other relevant outcomes, including the quality of life (QOL) score, pulmonary function test and the incidence of adverse event.

ELIGIBILITY:
Inclusion Criteria:

* Patients are suitable for inclusion in the study when they are 18 years or older diagnosed with COPD C group and bronchiectasis.

Exclusion Criteria:

* active tuberculosis
* severe respiratory disease (such as Lung cancer, ARDS, pulmonary encephalopathy, respiratory failure)
* uncontrollable diabetes
* hypersensitivity to any components of ICS/LABA or LAMA.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2017-09-15 (Actual); Primary Completion 2020-09-15 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
Acute exacerbation | 12 months
  The times of acute exacerbation during the trial.

SECONDARY OUTCOMES:
Number of patients with adverse events | 12 months
  All of the adverse events occurred in the processing of the trial,especially the prevalence of pneumonia.
FEV1 | 12 months
  Forced Expiratory Volume in one second
FVC | 12 months
  Forced Vital Capacity
FEV1/FVC | 12 months
  Pulmonary function test
SGRQ | 12 months
  St. George's Respiratory Questionnaire
LCQ | 12 months
  The Leicester Cough Questionnaire
CAT | 12 months
  COPD Assessment Test
mMRC | 12 months
  Modified Medical Research Council Dyspnea Scale

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Fu Xu, Principal Investigator — Shanghai Pulmonary Hospital , Tongji University
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Result] Oba Y, Lone NA. Comparative efficacy of inhaled corticosteroid and long-acting beta agonist combinations in preventing COPD exacerbations: a Bayesian network meta-analysis. Int J Chron Obstruct Pulmon Dis. 2014 May 12;9:469-79. doi: 10.2147/COPD.S48492. eCollection 2014. PMID 24872685
- [Result] Kew KM, Dias S, Cates CJ. Long-acting inhaled therapy (beta-agonists, anticholinergics and steroids) for COPD: a network meta-analysis. Cochrane Database Syst Rev. 2014 Mar 26;2014(3):CD010844. doi: 10.1002/14651858.CD010844.pub2. PMID 24671923
- [Result] Manoharan A, Short PM, Anderson WJ, Lipworth BJ. Impact of long-acting bronchodilators and exposure to inhaled corticosteroids on mortality in COPD: a real-life retrospective cohort study. Lung. 2014 Oct;192(5):649-52. doi: 10.1007/s00408-014-9611-8. Epub 2014 Jun 22. PMID 24952426